CLINICAL TRIAL: NCT07011537
Title: The Hinge Health and ENSO Back Pain Study: Prospective, Open-label, Randomized Superiority Trial of a Digital Health Program and High Frequency Impulse Therapy (HFIT) Versus Standard of Care in Treatment of Chronic Low Back Pain
Brief Title: Examining the Impact of a Digital Health Program and TENS Device for Patients With Chronic Low Back Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hinge Health, Inc (Industry)
Collaborators: Optum, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1389625
Record Dates: First submitted 2025-06-05; First posted 2025-06-08 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Back Pain Lower Back Chronic; Chronic Pain; Musculoskeletal Pain
Keywords: Chronic Pain; Chronic Back Pain; Chronic Lower Back Pain; Mechanical Back Pain; Degenerative Disc Disease; Degenerative Arthritis; Disc Compression
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain; Intervertebral Disc Degeneration; Osteoarthritis | interventions — Masks; Transcutaneous Electric Nerve Stimulation; Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hinge Health + Enso (Experimental): The intervention group will receive access to the Hinge Health program and an Enso device.
  Interventions: Behavioral: Digital Musculoskeletal (MSK) Program; Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Standard of Care (Other): The control group will continue to receive access to traditional medical care for their musculoskeletal needs through their healthcare provider.
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Behavioral: Digital Musculoskeletal (MSK) Program — Hinge Health is a digital MSK program to help participants manage chronic MSK pain through offering exercise therapy sessions, educational articles, and personal health coaching. Hinge Health delivers exercise therapy sessions and education through "playlists" accessed through the program app. Each playlist consists of three to seven exercises specific to the body region(s) the participant experiences pain in. Animations and videos, while paired with sensors and computer vision, demonstrate how to perform exercises, the number of repetitions for each exercise, and how long to hold positions. Playlists present more challenging exercises and/or more repetitions as participants progress further along in the program. After participants complete the exercises, the playlist delivers educational articles and resources focused on MSK pain-related topics, including lifestyle changes, pain neuroscience, and social support.
  Other Names: Hinge Health Program
  Arms: Hinge Health + Enso
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — The Enso is a strong complement/enhancement to the Hinge Health program, as it helps users to better manage their pain in order to work through their exercise sessions in the program. The Enso device is not intended to be a stand-alone solution; it provides pain relief, but exercise therapy provides important long-term benefits. Participants will use the digital MSK program (Hinge Health) in combination with a pain management device (Enso).
  Other Names: ENSO Device
  Arms: Hinge Health + Enso
Other: Standard of Care (SOC) — The control group will continue to receive the access to traditional medical care for their MSK needs through their healthcare provider. Upon study completion, control group members who complete all follow-up surveys will receive Hinge Health membership and an Enso device for free for 12 months, starting at the conclusion of their participation in the study.
  Other Names: Traditional Medical Care
  Arms: Standard of Care

SUMMARY:
The goal of this study is to examine the extent to which Hinge Health, a digital musculoskeletal program, and Enso, a wearable pain relief device, have clinically significant impact on the pain, function, and health care use among patients undergoing non-imperative care for chronic lower back pain.

DETAILED DESCRIPTION:
Digital health approaches are a way to deliver conservative therapy through interactive methods. These approaches may expand access to care due to the convenience of digital health, as participants can access care services at all hours and locations. Research has shown that participants of digital health programs show significant improvements in pain.

Hinge Health is a digital musculoskeletal (MSK) program that aims to help people manage their MSK pain through exercise, education, and personal coaching. In previous research, Hinge Health has shown improvements in pain, functional, and health care use outcomes. Enso is a portable device for the treatment of chronic and acute types of MSK pain. The electrical pulses delivered by Enso incorporate neuromodulation at high frequency (0.1 to 10 MHz) in addition to the low frequency (0 to 1 KHz) pulses transmitted by more traditional transcutaneous electrical nerve stimulation (TENS) units. The result is a unique mechanism of action compared to the paresthesia resulting from the electrical pulses delivered by traditional TENS devices. Furthermore, Enso has shown promising clinical outcomes in a small, pilot RCT.

While the pilot study provided preliminary results demonstrating clinical improvements in the short term, there is a need for evidence about medium to long term outcomes, impact on mood, and the effect on healthcare utilization. Therefore, the purpose of this study is to examine the extent to which Hinge Health, with Enso, have clinically significant impact on the pain, function, and health care use among patients undergoing non-imperative care for their chronic lower back pain in the medium and long term.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* United Healthcare (UHC) is primary health plan
* Mechanical (myofascial), axial back pain (focused around the spine)
* Experiencing pain primarily in the low back area
* Radicular component of pain has minimal effect on functionality, medication, quality of life
* Experiencing low back pain for at least 3 months
* Subject able to understand and provide informed consent
* Comfortable and willing to accept random assignment to one of two study conditions (intervention or standard care condition)
* Has an email account

Exclusion Criteria:

* Patients that do not own or have access to a smartphone or tablet
* Has spinal instability, joint instability, or grade 2 or greater spondylolisthesis with instability
* Primary symptoms due to spinal stenosis as evidenced by pseudoclaudication, leg weakness or numbness
* Source of back pain related to an acute nerve impingement
* Diagnosis of cancer/malignant tumors in the last 5 years
* Source of back pain is an infection
* History of spinal fusion surgery
* Has a cardiac pacemaker, implanted defibrillator, spinal cord stimulator, pain pump, or any other implanted electronic device
* Has had myocardial infarction within the past 6 months
* Has had a coronary stent in the past 3 months
* Has radicular pain symptoms that affect functionality, quality of life or medication intake
* Has undergone surgery to solve pain related to the study indication in the past 12 months
* Is scheduled for upcoming surgery to solve pain related to the study indication
* History of opioid or drug use, or excessive alcohol use (excessive alcohol use defined as greater than 3 drinks a day on average), per investigator discretion
* History of rheumatological or other inflammatory conditions such as rheumatoid arthritis, systemic lupus, erythematosus, etc.
* Any psychiatric condition that may interfere with the study assessments or prevent the subject from complying with the requirements of the protocol, in investigator's judgment
* Pregnant women (as determined by self-report)
* Has a heart condition that limits the ability to do mild exercise due to symptoms such as fatigue, palpitations, shortness of breath, or chest pain
* Has any health condition that limits the ability to do light-intensity exercise such as slow walking or light household chores
* Diagnosed with dementia or a similar memory disorder
* Has had a fall in the past three months
* Unable to move from sitting to standing without help from another person
* Unable to stand without assistance from another person or device
* Any other disease, condition, or habit(s) that in the opinion of the Principal Investigator would interfere with study compliance or adversely affect study outcomes
* Inability to complete data collection as required
* No secondary/coinsurance or plans to change insurance from UHC in the next 3 months
* Patients who were recommended spine surgery from a spine surgeon in the 3 months prior to the index month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Pain | Baseline, 2, 6, and 12 weeks
  Pain in the last 24 hours and at its worst in the last week will be measured via a Numerical Pain Rating Score (NPRS) with 0 indicating no pain and 100 indicating worst imaginable pain.
Change in Pain | Baseline, 2, 6, and 12 weeks
  In addition to the NPRS, Patient Global Impression of Change (PGIC) in pain will be collected based on the response to the question, "Compared to before starting this study, how would you rate your back pain now?" (Much Worse, Worse, A Little Worse, No Change, A Little Better, Better, Much Better), on a 0 to 7 scale.

SECONDARY OUTCOMES:
Function | Baseline, 2, 6, and 12 weeks
  Function will be measured using the Roland Morris Disability Questionnaire 11-item scale (RMDQ-11), ranging from 0 to 11. Change will be measured as baseline score minus follow-up score.
Depression | Baseline, 2, 6, and 12 weeks
  Depression symptoms will be measured with the Patient Health Questionnaire 8-item scale (PHQ-8), ranging from 0 to 24. Change will be measured as baseline score minus follow-up score.
Anxiety | Baseline, 2, 6, and 12 weeks
  Anxiety symptoms will be measured with the Generalized Anxiety Disorder 7-item scale (GAD-7), ranging from 0 to 21. Change will be measured as baseline score minus follow-up score.

OTHER OUTCOMES:
Healthcare Utilization and Costs | Baseline, 12 months
  Healthcare utilization and cost data will be come from administrative claims data and prescription history. These data will be collected for the intervention and control groups and will include 12 months of retrospective healthcare utilization claims records.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Cohen, MD, FACP, Principal Investigator — Optum, Inc.; Jeff Krauss, MD, Principal Investigator — Hinge Health; Cynthia Castro Sweet, PhD, Principal Investigator — Hinge Health
Locations (1):
- Optum Labs, Eden Prairie, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No